CLINICAL TRIAL: NCT03720834
Title: What is the Numerical Translation of Verbal Probability Expressions Used by Patients and Doctors in the Context of Communication of Peri-operative Risk?
Brief Title: Verbal Probability Expressions in Peri-operative Risk
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH20393
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Surgery--Complications; Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Questionnaire on risk perception
- Clinicians: Questionnaire on risk perception

SUMMARY:
Before having an operation doctors use expressions such as high risk, or low risk to describe the chance of complications occurring. Complications include things such as strokes and heart attacks and even death. It is thought that using words like this, instead of percentages makes it easier for patients to understand their level of risk. It is also often hard for a doctor to give a patient an exact percentage.

It is important that patients have a good understanding about their level of risk associated with an operation so they can make informed decisions about whether to go ahead with it. This is an important part of taking consent before an operation.

The aim of this study is to assess whether using expressions such as high risk and low risk to communicate the chance of a complication occurring during an operation is useful.

Different patients may assign different meanings to these expressions. If it is found that patients interpret these expressions differently from how the doctor intended it would suggest that the way doctors communicate risk to patients should be reviewed.

Patients will be asked if they are willing to participate in the study and after giving consent they will complete a questionnaire. The questionnaire will list various expressions used by doctors to describe the chance of a complication occurring during an operation, such as high risk and low risk. Each participant will be asked to give a percentage for each of the expressions. The questionnaire will be completed by patients who are waiting to have an operation at the Royal Hallamshire Hospital.

DETAILED DESCRIPTION:
Shared decision-making is central to the consent process prior to surgery and anaesthesia. Verbal probability expressions are commonly used by clinicians to help describe the level of risk. Common examples of verbal probability expressions are shown below with the estimated numerical risk shown in parentheses:

* High risk (1:100)
* Moderate risk (1:100-1:1000)
* Low risk (1:1000-1:10 000)
* Standard risk (varies depending on patient/procedure etc.)
* Very low risk (1:10 000)
* Minimal risk (1:100 000)
* Negligible risk (1:1 000 000)

Verbal probability expressions are commonly used because they are perceived as being easier to understand than, for example, percentage risk, as this is affected by how numerate a patient is. Clinicians often prefer verbal probability expressions as they avoid assigning an exact percentage of risk; this is because risk prediction is an inexact science and from an individual patient perspective, risk of complications is often a dichotomous outcome - their individual experience will be either a 0% or 100% incidence of complications, depending on whether it happens to them or not. Percentage risk only really applies to large populations, not individual patients.

Shared decision-making is central to the consent process prior to surgery and anaesthesia. With pre-operative clinics, risk indices are often described according to Calman's verbal scale illustrated above (high, moderate, low, very low etc.). However, the actual level of harm that is perceived by the patient and clinician may differ, due a variety of factors, not least a lack of understanding of the underlying numerical concepts. In addition, the level of risk assigned to these by clinicians and the level perceived by patients may differ. For example, a clinician may view a 20% probability of a complication after cancer surgery is high-risk, when compared to their own experience of the procedure; the patient who is living with the disease may see this as a low-risk, given their individual perception of the disease.

This study aims to investigate this and to see if verbal probability expressions are still useful for communication of pre-operative risk. If the study finds large inter-individual variability between patients, then this would suggest that the use of verbal probability expressions in discussions should be reviewed. This may include the need for verbal probability expressions to be used in conjunction with a numerical estimate of risk, or for the terms used (high-risk, low-risk) to be revised. The results of this study may have significant implications at national level in terms of the consent process for surgical procedures.

After gaining consent, a questionnaire with various verbal probability expressions will be completed by clinicians and patients. Each participant will be asked to assign a percentage of likelihood (i.e. a numerical translation) of an adverse outcome according to each verbal probability expression. For example, one patient may perceive the phrase 'high-risk" as an incidence risk in excess of 50%, whilst another may perceive the risk to be 20%.

A researcher will be available to answer any questions will occur during the completion of the questionnaire.

The study is observational.

The numerical translation of different verbal probability expressions will be displayed graphically to illustrate variation (if any). For example, if the phrase 'high-risk" is perceived by patients as a percentage risk ranging from 20-70%, whilst anaesthetists and surgeons perceive 'high-risk' as 10-20%, then this particular verbal probability expression would be of limited value.

We will use ANOVA to analyse if there is any difference in the level risk assigned to different verbal probability expressions by patients and anaesthetists (after testing for normality of data distribution). For example, do patients recognise a meaningful difference between low and minimal risk?

Regression analyses will also be undertaken to determine if any patient factors alter the perception of risk. This will include: sex; calculated Surgical Outcome Risk Tool score; cancer vs. non-cancer surgery; ethnicity; and surgical speciality.

ELIGIBILITY:
Inclusion Criteria:

* Any patient due to undergo surgery who attends pre-operative assessment clinic

Exclusion Criteria:

* Inability to speak/read English; inability to provide own consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Surgical population
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
To determine the perceived peri-operative risk (as a percentage incidence) associated with a variety of verbal probability expressions in patients awaiting surgery. | Day 0
  Percentage risk assigned to verbal risk descriptors

SECONDARY OUTCOMES:
To determine the implied patient peri-operative risk (as a percentage incidence) associated with a variety of verbal probability expressions that are used by clinicians in the pre-operative setting. | Day 0
  Percentage risk assigned to verbal risk descriptors
To determine the level of correlation between clinicians and patient perception of risk when verbal probability expressions are used. | Day 0
  Percentage risk assigned to verbal risk descriptors
To investigate the impact of patient sex, surgical speciality, presence of carcinoma, and calculated risk of surgery on patient perception of risk when verbal probability expressions are used. | Day 0
  Logistic regression

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No